CLINICAL TRIAL: NCT02124551
Title: Comparing PVI Measurements at Different Sensing Locations
Brief Title: Comparing Pleth Variability Index (PVI) Measurements at Different Sensing Locations
Status: Completed | Type: Observational
Sponsor: University of California, Irvine (Other)
Collaborators: Masimo Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: UCIANES05
Record Dates: First submitted 2014-04-24; First posted 2014-04-28 (Estimated); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Fluid Imbalance
Keywords: Goal-directed fluid therapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to assess the suitability of the ear and forehead as a better site for measure of fluid responsiveness.

DETAILED DESCRIPTION:
The aim of this study is to compare Pleth Variability Index (PVI) measurements at different sensor locations in respect to signal quality, sensor fit to site location and fluid responsiveness. PVI will be measured at 3 different sensor sites: the fingers, ear lobes and forehead. The ability to predict fluid responsiveness will be analyzed using cardiac output as the reference value.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Undergo any type of surgeries under general anesthesia in UCI Medical Center
* Mechanically ventilated during surgery
* Arterial line placement is preferred but not required
* Agree to sign the consent and HIPAA forms

Exclusion Criteria:

* Less than 18 years of age
* Pregnant women
* Refused to sign the consent and HIPAA forms
* Receive vasoactive medication prior to surgery
* Has these conditions: hypotension, hypothyroidism, moderate or poorly controlled hypertension, chronic poorly-controlled diabetes, heart failure patients, and patients with active airway flow obstruction, left ventricular dysfunction, intra-cardiac shunts, right ventricular dysfunction, atrial fibrillation, arrhythmias
* patients with surgeries at or around site of sensor placement
* Subject has skin abnormalities affecting the digits such as psoriasis, eczema, angioma, scar tissue, burn, fungal infection, substantial skin breakdown, nail polish or acrylic nails that would prevent monitoring of SpO2 levels during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be patients who undergo any form of surgery, where he/she is mechanically ventilated, preferably cases that require arterial line placement, use of cardiac output measurement, and where fluid administration will occur perioperatively.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2014-04; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
PVI measurement of fluid responsiveness | Intra-operative
  The primary outcome is to test the ability of PVI recorded at the finger and at the ear to predict fluid responsiveness.

CONTACTS AND LOCATIONS:
Overall Officials: Maxime Cannesson, PhD, Principal Investigator — UC Irvine
Locations (1):
- University of California, Irvine Medical Center, Orange, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cannesson M, Besnard C, Durand PG, Bohe J, Jacques D. Relation between respiratory variations in pulse oximetry plethysmographic waveform amplitude and arterial pulse pressure in ventilated patients. Crit Care. 2005 Oct 5;9(5):R562-8. doi: 10.1186/cc3799. Epub 2005 Aug 23. PMID 16277719
- [Background] Feissel M, Teboul JL, Merlani P, Badie J, Faller JP, Bendjelid K. Plethysmographic dynamic indices predict fluid responsiveness in septic ventilated patients. Intensive Care Med. 2007 Jun;33(6):993-9. doi: 10.1007/s00134-007-0602-6. Epub 2007 Mar 29. PMID 17393139
- [Background] Cannesson M, Attof Y, Rosamel P, Desebbe O, Joseph P, Metton O, Bastien O, Lehot JJ. Respiratory variations in pulse oximetry plethysmographic waveform amplitude to predict fluid responsiveness in the operating room. Anesthesiology. 2007 Jun;106(6):1105-11. doi: 10.1097/01.anes.0000267593.72744.20. PMID 17525584
- [Background] Cannesson M, Delannoy B, Morand A, Rosamel P, Attof Y, Bastien O, Lehot JJ. Does the Pleth variability index indicate the respiratory-induced variation in the plethysmogram and arterial pressure waveforms? Anesth Analg. 2008 Apr;106(4):1189-94, table of contents. doi: 10.1213/ane.0b013e318167ab1f. PMID 18349191
- [Background] Hood JA, Wilson RJ. Pleth variability index to predict fluid responsiveness in colorectal surgery. Anesth Analg. 2011 Nov;113(5):1058-63. doi: 10.1213/ANE.0b013e31822c10cd. Epub 2011 Sep 30. PMID 21965349
- [Background] Shelley KH, Jablonka DH, Awad AA, Stout RG, Rezkanna H, Silverman DG. What is the best site for measuring the effect of ventilation on the pulse oximeter waveform? Anesth Analg. 2006 Aug;103(2):372-7, table of contents. doi: 10.1213/01.ane.0000222477.67637.17. PMID 16861419
- [Background] Cannesson M, Desebbe O, Rosamel P, Delannoy B, Robin J, Bastien O, Lehot JJ. Pleth variability index to monitor the respiratory variations in the pulse oximeter plethysmographic waveform amplitude and predict fluid responsiveness in the operating theatre. Br J Anaesth. 2008 Aug;101(2):200-6. doi: 10.1093/bja/aen133. Epub 2008 Jun 2. PMID 18522935